CLINICAL TRIAL: NCT02153606
Title: Glycerin Suppositories Used Prophylactically in Premature Infants (SUPP): a Pilot Randomized Placebo-controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: McMaster Surgical Associates (Other); Hamilton Health Sciences Corporation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Walton-MSA14-GlycerinSupp
Record Dates: First submitted 2014-05-23; First posted 2014-06-03 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Feeding Intolerance in Premature Infants
Keywords: Glycerin Suppositories; Enteral Nutrition; Enterocolitis, Necrotizing; Infant, Premature; Meconium
MeSH Terms: conditions — Enterocolitis, Necrotizing; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Glycerin Suppository (Active Comparator)
  Interventions: Drug: Glycerin Suppository
- Sham Suppository (Sham Comparator)
  Interventions: Other: Sham Suppository

INTERVENTIONS:
Drug: Glycerin Suppository — The treatment intervention will be a 250 mg glycerin suppository placed in the rectum once daily starting 48-72 hours after birth.
  Arms: Glycerin Suppository
Other: Sham Suppository — Sham suppositories will be created by placing a 250 mg glycerin suppository in the diaper once daily starting 48-72 hours after birth. This intervention works as a non-invasive placebo to maintain blinding.
  Arms: Sham Suppository

SUMMARY:
All premature babies have problems with feeding and nutrition. Some can develop a life-threatening bowel infection necrotizing enterocolitis. This can result in the need for emergency surgery, loss of bowel, lifelong feeding problems, and death. Giving premature babies glycerin suppositories may be one way to stimulate the digestive tract and help prevent these problems. To see if this treatment works, the investigators need to study hundreds of premature babies in a large trial involving multiple hospitals. The purpose of this project is to carry out a small study first and make sure that the larger trial is feasible. The investigators will invite approximately 30 premature babies from the Neonatal Intensive Care Unit at McMaster University Medical Centre to participate in this study over a 6-month period. The investigators will focus on feasibility issues, including cost, safety, and rate of participation. This will allow us to rigorously test our study protocol and lay the groundwork for the larger study involving multiple hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age 24-32 weeks OR
* Birth weight 500-1500 grams

Exclusion Criteria:

* Congenital gastrointestinal anomalies
* Surgery within 48 hours of birth
* Culture-proven sepsis*
* Vasopressors within 6 hours of first intervention
* Nitric oxide
* Duct-dependent congenital heart defect requiring prostaglandins
* Suspected coagulopathy (mucosal bleeding from any orifice)
* Confirmed coagulopathy (any one of the following):
* International Normalized Ratio greater than 1.4
* Partial Thromboplastin Time greater than 39 seconds
* Fibrinogen less than 1.00 grams/liter
* Thrombocytopenia (platelet count less than 100 x 10^9/liter)**
* Neutropenia (absolute neutrophil count less than 0.5 x 10^9/liter)
* Complete meconium evacuation (2 normal bowel movements) within 48 hours of life
* Parent or legal guardian unable to understand English

Note:

* C-reactive protein is not an exclusion criteria

** Indomethacin alone is not an exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Days to full enteral feeding (150 ml/kg/day) | Up to 4 months

SECONDARY OUTCOMES:
Feeding volume on day 14 of life (ml/kg/day) | 14 days
Days to complete meconium evacuation | Up to 4 months
  Number of days to complete meconium evacuation (defined as two normal bowel movements free of meconium staining).
Compliance with treatment regimen | Up to 4 months
Days of parenteral nutrition | Up to 4 months
Necrotizing enterocolitis | Up to 4 months
Culture-proven line sepsis | Up to 4 months
Mortality | Up to 4 months

OTHER OUTCOMES:
Recruitment rate | 6 months
  Percentage of eligible infants randomized
Completion rate | 6 months
  Percentage of randomized infants reaching full enteral feeds
Treatment-related adverse events | Up to 4 months
  Rectal perforation, rectal bleeding, and/or anal fissure
Cost | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: J M Walton, M.D., Principal Investigator — McMaster University
Locations (1):
- McMaster University Medical Centre, Hamilton, Ontario, Canada

REFERENCES:
- [Derived] Livingston MH, Zequeira J, Blinder H, Pemberton J, Williams C, Walton JM. Glycerin suppositories used prophylactically in premature infants (SUPP) trial: a study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2015 Aug 25;1:31. doi: 10.1186/s40814-015-0024-0. eCollection 2015. PMID 27965809